CLINICAL TRIAL: NCT00318968
Title: Development of an Algorithm for Identification of Responders to Short Term Treatment With Esomeprazole (Nexium) in Primary Care
Brief Title: Nexium RESPONSE Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: D9612L00076; RESPONSE
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: GERD
Keywords: Acid Reflux; Nexium; Esomeprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
The primary purpose of the study is to develop, and test, an algorithm for identification of responders to empirical esomeprazole treatment in general practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending general practice due to symptoms suggestive of acid related disease and, according to normal routine, the GP would prescribe an acid-inhibiting agent

Exclusion Criteria:

* Alarm symptoms
* Pregnancy
* Contraindications to Nexium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-05; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the patient's key complaint. A patient whose key complaint has been absent for the last 24 hour of the treatment period (2 weeks +/- 2 days) is defined as a PPI responder.

SECONDARY OUTCOMES:
To evaluate the response rate (absence of the key complaint for the last 3 days of the treatment period (2 weeks +/- 2 days)).

CONTACTS AND LOCATIONS:
Overall Officials: Villy Meineche Schmidt, MD, Principal Investigator — Charlottenlund Research Site; Stig Waldorff, MD, Study Director — AstraZeneca, Denmark
Locations (38):
- Denmark (38):
  - Research Site, Aabenraa
  - Research Site, Aalborg
  - Research Site, Albek
  - Research Site, Ans
  - Research Site, Arhus C
  - Research Site, Bagsværd
  - Research Site, Birkerød
  - Research Site, Brønshøj
  - Research Site, Farum
  - Research Site, Fredericia
  - Research Site, Frederikshavn
  - Research Site, Frederikssund
  - Research Site, Gråsten
  - Research Site, Haslev
  - Research Site, Herning
  - Research Site, Hinnerup
  - Research Site, Karlslunde
  - Research Site, Kerteminde
  - Research Site, Kobenhavn K
  - Research Site, Kolding
  - Research Site, Løsning
  - Research Site, Middelfart
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Randers
  - Research Site, Roskilde
  - Research Site, Rungsted Kyst
  - Research Site, Rødovre Municipality
  - Research Site, Saltum
  - Research Site, SEBY
  - Research Site, Sindal
  - Research Site, Solrød Strand
  - Research Site, Svendborg
  - Research Site, Tåstrup
  - Research Site, Tønder
  - Research Site, Ullerslev
  - Research Site, Viborg
  - Research Site, Viby J

REFERENCES:
- [Derived] Bytzer P, Langkilde LK, Christensen E, Meineche-Schmidt V. Work productivity improvement after acid suppression in patients with uninvestigated dyspepsia. Dan Med J. 2012 Jul;59(7):A4461. PMID 22759841
- [Derived] Meineche-Schmidt V, Christensen E, Bytzer P. Randomised clinical trial: identification of responders to short-term treatment with esomeprazole for dyspepsia in primary care - a randomised, placebo-controlled study. Aliment Pharmacol Ther. 2011 Jan;33(1):41-9. doi: 10.1111/j.1365-2036.2010.04501.x. Epub 2010 Oct 29. PMID 21083590